CLINICAL TRIAL: NCT00848601
Title: Safety Study to Determine the Maximum Tolerated Dose, Pharmacokinetics and Pharmacodynamics of SGI-1776, a PIM Kinase Inhibitor, in Subjects With Hormone and Docetaxel Refractory Prostate Cancer and Relapsed/Refractory Non Hodgkin's Lymphoma
Brief Title: Safety of SGI-1776, A PIM Kinase Inhibitor in Refractory Prostate Cancer and Relapsed/Refractory Non Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The dose limiting toxicity of cardiac QTc prolongation was identifiedin the phase 1 study in patients with refractory prostate and lymphoma
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SGI-1776-01
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer; Non-Hodgkins Lymphoma
Keywords: SGI-1776; PIM; Hormone & Docetaxel refractory Prostate Cancer; Refractory non-Hodgkin's Lymphoma
MeSH Terms: conditions — Prostatic Neoplasms; Lymphoma, Non-Hodgkin | interventions — SGI 1776

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SGI-1776 — Starting dose 100 mg (total daily dose) administer as 50 mg every 12 hours for 14 days of a 21-day cycle, dose escalation in successive cohorts until progression or toxicity develops

SUMMARY:
Patients with hormone and docetaxel refractory prostate cancer or relapsed/refractory non-Hodgkin's lymphoma for which no available standard therapy or therapy which may provide clinical benefit is available will be enrolled. Primary objectives: estimate the maximum tolerated dose and dose-limiting toxicities. Secondary objectives: Response rate, pharmacokinetic and pharmacodynamic profiles, Prostate Specific Antigen response and renal elimination.

ELIGIBILITY:
General

Inclusion Criteria:

1. Read, understand and sign the IRB- or IEC-approved ICF confirming his or her willingness to participate in this trial.
2. At least 18 years old.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
4. Adequate bone marrow function; normal renal and hepatic function, normal cardiac function.
5. Normal cardiac function in the opinion of the investigator and supported by LVEF 50% or greater on the screening echocardiogram (or MUGA), no significant abnormalities on the screening ECG (eg, left bundle branch block, III degree AV block, acute myocardial infarction, Wolff-Parkinson-White syndrome or QTc interval ≥ 450 msec) and no history of additional risk factors for torsades de pointes (eg, heart failure, hypokalemia or family history of Long QT Syndrome).

Exclusion Criteria:

1. Active secondary malignancy or history of other malignancy within the last two years except non-melanoma skin cancers or cervical carcinoma in situ.
2. History of significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure and/or myocardial infarction or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
3. Received any anticancer agent(s) within the past 3 weeks, including investigational agents, chemotherapy (6 weeks for nitrosoureas or mitomycin), immunotherapy, biologic or marketed or investigational tyrosine kinase inhibitors.
4. Received prior radiation therapy within the past 4 weeks or received irradiation of ≥ 25% of their bone marrow reserve.
5. Any serious, uncontrolled active infection that requires systemic treatment or known infection with HIV, HCV or HBV.
6. Symptomatic CNS metastases or lesions for which treatment is required.

Prostate Cancer

Inclusion Criteria:

1. Males with histologically confirmed adenocarcinoma of the prostate, which is now metastatic (e.g., any T, any N, M1a-c)based on bone scan, CT scan, or MRI scan. Demonstrated evidence of progressive disease despite androgen deprivation (androgen ablation or surgical castration), anti-androgen withdrawal and progression of disease after docetaxel-based therapy.
2. Demonstrated evidence of progressive disease despite androgen deprivation (androgen ablation or surgical castration), anti-androgen withdrawal and progression of disease after docetaxel-based therapy.

   • Greater than 25% increase in 3 consecutive tests (PSA 1 < PSA 2 < PSA 3), each PSA value separated by at least 1 week
3. Serum testosterone level ≤ 50 ng/dL post orchiectomy or while maintained on continuous or intermittent medical androgen suppression with a LHRH agonist or antagonist.
4. At least 4 weeks since prior flutamide, megestrol, ketoconazole, aminoglutethimide; and at least 6 weeks since prior bicalutamide or nilutamide.
5. Systemic corticosteroids discontinued within two weeks of dosing, except low dose regimens which may continue if unchanged
6. Strontium-89 or Samarium-153 must have been completed at least 8 weeks prior to the first dose of therapy and recovered from all treatment-related toxicities.

Exclusion Criteria:

1. Must not be receiving concurrent anti-androgen hormonal therapy for hormone refractory prostate cancer.

Non-Hodgkin's Lymphoma

Inclusion Criteria:

1. Histologically proven relapsed or refractory non-Hodgkin's lymphoma subjects for which there is no available standard therapy or therapy which may provide clinical benefit.
2. Measurable disease (at least 1 lesion ≥ 1.5 cm).

Exclusion Criteria:

1. Bulky disease by CT, defined as any single mass >10 cm in its greatest diameter.
2. Systemic corticosteroids within 2 weeks, except low dose regimens which may continue if unchanged.
3. Received any radiopharmaceutical therapy within the past six weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
MTD & DLT | July 2011

SECONDARY OUTCOMES:
Response rate, pharmacokinetics, PSA response, renal elimination and pharmacodynamic effects on biomarker modulation. | July 2011

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - UCLA, Los Angeles, California
  - Cancer Therapy Research Center, San Antonio, Texas
- Royal Marsden Hospital, Sutton, England, United Kingdom